CLINICAL TRIAL: NCT06176729
Title: A Prospective Phase II Study of Polatuzumab, Rituximab, and Lenalidomide(Pola-R2) in Newly-diagnosed Non-fit Elderly DLBCL Patients
Brief Title: Pola-R2 in Newly Diagnosed Non-fit Elderly DLBCL Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yan Zhang, MD (Other)
Collaborators: Peking University Third Hospital (Other); Peking University First Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Yan Zhang, MD, associate director of department of hematology, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-PUMCH-A-194
Record Dates: First submitted 2023-12-05; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Pola-R2 regimen Drug: Polatuzumab Vedotin, Rituximab, Lenalidomide polatuzumab vedotin 1.8 mg/kg ivgtt D1, rituximab375 mg/m2 ivgtt D1, lenalidomide 25mg po D1-14, one cycle every 21 days
  Interventions: Drug: Polatuzumab Vedotin, Rituximab, Lenalidomide

INTERVENTIONS:
Drug: Polatuzumab Vedotin, Rituximab, Lenalidomide — polatuzumab vedotin 1.8 mg/kg ivgtt D1, rituximab375 mg/m2 ivgtt D1, lenalidomide 25mg po D1-14, one cycle every 21 days

SUMMARY:
This is a prospective, single-arm, phase II study, and the purpose of this study is to evaluate the efficacy and safety of Pola-R2 regimen in newly diagnosed elderly diffuse large B cell lymphoma classified into un-fit or frail group by comprehensive geriatric assessment(CGA).

DETAILED DESCRIPTION:
In this prospective study, all the eligible patients will be given Pola-R2 regimen(polatuzumab vedotin 1.8 mg/kg ivgtt D1, rituximab375 mg/m2 ivgtt D1, lenalidomide 25mg po D1-14, one cycle every 21 days). An interim evaluation will be performed after 4 cycles, the patients who achieve CR or PR will receive another 4 cycles of Pola-R2.

The patients with stable disease (SD) or progressed disease (PD) will withdraw from the trial and receive salvage regimens.

ELIGIBILITY:
Inclusion Criteria:

* The patient volunteered to participate in the study and signed the Informed Consent
* Histopathologically confirmed DLBCL and treatment naive(corticosteroids alone is not considered as a line of treatment)
* Age≥ 70 years old, and was un-fit or frail according to comprehensive geriatric assessment
* Adequate organ function and adequate bone marrow reserve

Exclusion Criteria:

* Coexisting malignancy other than lymphoma
* Active HBV infection
* Any instability of systemic disease, including but not limited to active infection (except local infection), severe cardiac, liver, kidney, or metabolic disease need therapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-10-24 (Estimated); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | evaluated every 3 months，up to 24 months
  proportion of patients achieving complete remission

SECONDARY OUTCOMES:
overall remission rate | evaluated every 3 months，up to 24 months
  proportion of patients achieving at least partial remission
2 year progression-free survival rate | 2 years after last patient included
  time from treatment to the time of disease progression or death of any reason
2 year overall survival rate | 2 years after last patient included
  time from treatment to the time of death of any reason
any adverse event occurred during this study | 2 years after last patient included
  safety

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No